CLINICAL TRIAL: NCT02956148
Title: Follow-up Measurement of Brain Phosphodiesterase 10 A (PDE10A) Enzyme Levels in Huntington´s Disease Gene Expansion Carriers, 18 to 28 Months After Initial Positron Emission Tomography (PET) Measurement in CHDIKI1201/PET-HD-PDE10A (NCT02061722)
Brief Title: Follow-up Measurement of Brain PDE10A Enzyme Levels in Huntington´s Disease Gene Expansion Carriers
Acronym: LONGPDE10
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: CHDI Foundation, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHDIKI1401
Record Dates: First submitted 2016-03-11; First posted 2016-11-07 (Estimated); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Huntington's Disease
MeSH Terms: conditions — Huntington Disease | interventions — 2-(2-(3-(4-(2-fluoroethoxy)phenyl)-7-methyl-4-oxo-3,4-dihydroquinazolin-2-yl)ethyl)-4-isopropoxyisoindoline-1,3-dione

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radioligand [18F]MNI-659 (Experimental): All subjects will receive a single intravenous dose of the radioligand [18F]MNI-659 (investigational medicinal product [IMP]) and undergo PET imaging.
  The radioligand [18F]MNI-659 will be administered at a dose of less than 5 micrograms, i.e. within the micro dosing concept, and no pharmacological effects are expected.
  The injected radioactivity of [18F]MNI-659 will be 185 MBq/70 kg of body weight ± 10%.
  Interventions: Radiation: Radioligand [18F]MNI-659

INTERVENTIONS:
Radiation: Radioligand [18F]MNI-659 — The effective radiation dose for the injection of [18F]MNI-659 is approximately 5.6 mSv (approximately 2 years of background radiation in Sweden) for an average person weighing 70 kg.

SUMMARY:
The aim of this study is to measure longitudinally the availability of the PDE10A enzyme in HDGECs using the radioligand [18F]MNI-659. The study will be a follow-up, examining HDGECs from the CHDIKI1201/PET-HD-PDE10A (NCT02061722) study from 18 to 28 months after the initial PET measurement.

DETAILED DESCRIPTION:
The HDGECs will perform 2 study visits: Visit 1 (screening) and Visit 2 (PET analysis utilizing the radioligand [18F]MNI-659). There will also be 2 telephone follow ups; one after Visit 1 (telephone follow-up after screening) and one after Visit 2, (telephone follow-up after PET). Study visits and telephone follow-ups will take place during a maximum of 97 days.

ELIGIBILITY:
Inclusion Criteria:

* Have participated in and completed study CHDIKI1201/PET-HD-PDE10A and are capable of providing informed consent or have a legal representative authorized to give consent on their behalf.
* Otherwise healthy according to medical history, no co-morbidity of psychotic disorders, physical examination, vital signs and laboratory assessments
* Willing to travel to Stockholm (with a companion if requested) for PET examinations
* Suitable physically and psychologically to travel to Stockholm and undergo PET examinations, as judged by the recruiting Investigator with attention given to symptoms of chorea and anxiety
* Willing to comply with the use of adequate contraceptive measures

Exclusion Criteria:

* Any disease, condition or concomitant medications that significantly compromises the function of the body systems and that, in the opinion of the Investigator might interfere with the conduct of the study or the interpretation
* Regular use of any medication prohibited by this protocol (selective or non-selective PDE inhibitors), with the exception for erectile dysfunction medication, which may be temporarily discontinued prior to the PET measurement
* History of anaphylactoid or anaphylactic reactions to any allergen including drugs and contrast media
* History of other neurological condition (including brain surgery, intracranial hematoma, stroke/cerebrovascular disorders, epilepsy), co-morbidity of psychiatric disorders
* Clinically relevant findings in hematological, biochemical testing or 12-lead ECG as determined by the evaluating physician
* Female subjects who are breast-feeding or have a positive pregnancy test at screening or at Visit 2

Ages: 18 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-09-06 (Actual); Primary Completion 2017-10-05 (Actual); Study Completion 2017-10-05 (Actual)

PRIMARY OUTCOMES:
The longitudinal changes of PDE10A enzyme availability in the caudate, putamen, and globus pallidus of Huntington's Disease Gene Expansion Carriers by comparison of the follow-up and initial PET measurements. | The follow up PET measurement can be performed from 18 to 28 months after the initial PET measurement that was performed in the CHDIKI/PET-HD-PDE10A Study
  The HDGECs will perform 2 study visits; Visits 1 (screening) and Visit 2 (PET) and 2 telephone follow ups, one after Visit 1 (telephone follow-up after screening) and one after Visit 2, (telephone follow-up after PET) 18 to 28 months after the initial PET measurement conducted in the CHDIKI1201/PET-HD-PDE10A study. An individual subject's participation in this study will last for a maximum of 97 days

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Varrone, MD, PhD, Principal Investigator — Karolinska University Hospital; Cristina Sampaio, MD, PhD, Study Director — CHDI Foundation, Inc.
Locations (7):
- The Memory Clinic, Rigshopitalet, Copenhagen, Denmark
- Leiden University Medical Center, Department of Neurology, Leiden, Netherlands
- University of Oslo, Nevrologisk poliklinikk, Oslo, Norway
- Sweden (4):
  - Skane Universitetssjukhus Lund, Neurologiska kliniken, Lund
  - Karolinska Universitetssjukhus, Huddinge, Stockholm
  - Karolinska University Hospital, Stockholm
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No